CLINICAL TRIAL: NCT04831411
Title: Comparison of Early Whole Body Vibration and Progressive Resistance Training to Enhance Recovery After Fast-Track Total Knee Arthroplasty: A Randomized Comparative Study.
Brief Title: Comparison of Early Whole Body Vibration and Progressive Resistance Training in Fast-Track Total Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gökhan Bayrak, Director, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBV-PRE training after TKA
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Knee Arthropathy
Keywords: fast-track surgery; whole body vibration; progressive resistance training; total knee arthroplasty; rehabilitation
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration (Active Comparator): The training program will last 2 days a week and 6 weeks in total. Each session includes a warm-up, progressive whole-body vibration training and a cooling exercise. On the remaining days of the week, all patients will apply the standard exercise program, which includes simple home exercises, at home.
  Interventions: Procedure: Total Knee Arthroplasty; Other: Whole Body Vibration
- Progressive Resistance Training (Active Comparator): The training program will last 2 days a week and 6 weeks in total. Each session includes a warm-up, progressive resistance training and a cooling exercise. On the remaining days of the week, all patients will apply the standard exercise program, which includes simple home exercises, at home.
  Interventions: Procedure: Total Knee Arthroplasty; Other: Progressive Resistance Training

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — The extremities of patients admitted to the operating room to be applied TKA will be determined using a safe surgical Fast-Track recovery protocol. Patients will be operated by the same surgical team using the same technique. Spinal anaesthesia or general anaesthesia will be applied to the patients according to the evaluations of the anesthesiologists.
Other: Whole Body Vibration — Whole Body Vibration
  Arms: Whole Body Vibration
Other: Progressive Resistance Training — Progressive Resistance Training
  Arms: Progressive Resistance Training

SUMMARY:
Patients who have undergone total knee arthroplasty (TKA) with Fast-Track recovery protocol at the Department of Orthopedics and Traumatology at the Local University Hospital and meet the inclusion and exclusion criteria will constitute the study sample. The patients will be divided into 2 groups using the computerized randomization method in the post-operative 4th week; Whole Body Vibration Group and Progressive Resistance Exercise Group. The first evaluation of the participants will be made at the end of the post-operative 4th week. Final evaluations will be made at the end of the post-operative 10th week, following the 6-week training.

DETAILED DESCRIPTION:
Patients who have undergone total knee arthroplasty (TKA) with Fast-Track recovery protocol at the Department of Orthopedics and Traumatology at the Local University Hospital and meet the inclusion and exclusion criteria will constitute the study sample. The patients will be divided into 2 groups using the computerized randomization method in the post-operative 4th week; Whole Body Vibration Group and Progressive Resistance Exercise Group. The first evaluation of the participants will be made at the end of the post-operative 4th week. After 2 days and 6 weeks of training a week, final evaluations will be made at the end of the 10th postoperative week. Evaluations will include measures of impairment in body functions and structures, activity limitation measures, balance assessment, and quality of life assessments. Evaluations will be made by a blind researcher. The study will be started with a total of 28 patients, including 14 participants in both groups. The sample size was determined by performing a power analysis. The purpose of the study will be explained to the patients by the researcher and the patients who agree to participate in the planned study will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing unilateral TKA surgery due to knee OA,
* Being between the ages of 50-75,
* To be able to understand the verbal and written information given.

Exclusion Criteria:

* To undergo revision TKA surgery.
* Participating in any exercise or strengthening training within the last 3 months.
* Having undergone major surgery on the extremity to be operated on.
* Having a comorbid disease such as rheumatoid arthritis, cancer.
* Having a neurological disease that causes functional insufficiency.
* Having a diagnosed psychiatric disorder.
* Having received anaesthesia for any reason in the last 1 month.
* Regularly using hypnotics or anxiolytics.
* Having dementia.
* Having a hearing or vision impairment that cannot be corrected with a hearing aid or glasses.
* Being morbidly obese (Body mass index> 40 kg/m2).
* Having implanted pacemakers or defibrillators.
* Having dermatological problems affecting the thigh.
* Having a score above 3 in the American Society of Anesthesiologists classification score.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Balance | 6 weeks
  Kinesthetic Ability Trainer® (KAT Model TS 650) will be used to evaluate balance. Patients will use the lines on the platform to place their feet in the same place for each measurement. Patients will be informed that the cursor on the system interface indicating the location of the pressure centre should be moved as little as possible and kept close to the centre. The rates of pressure centre change will be recorded as a result of the balance score obtained after 30 seconds of measurements on bipedal feet. Measurements will be applied in 3 repetitions and their average will be recorded and recorded in the study.
Quadriceps muscle strength | 6 weeks
  A handheld dynamometer (Commander Muscle Tester, JTech, USA) will be used for quadriceps muscle strength measurement. Patients will be seated on the treatment table with their hips and knees in 90 ° flexion with their feet hanging down. In this position, the hands will be on crossed shoulders and the use of bodyweight will be prevented. During the measurements, verbal guidance will be given to the patients in order to achieve maximum effort. Measurements will be made from the distal anterior face of the tibia with 3 consecutive maximum isometric contractions. The average of the measurement values will be recorded as a score.

SECONDARY OUTCOMES:
Pain assesment | 6 weeks
  Pain will be assessed by the Visual Pain Scale (pain perceived during rest, sleep and walking).
Western Ontario and McMaster Universities Osteoarthritis Index score | 6 weeks
  Western Ontario and McMaster Universities Osteoarthritis Index score is a patient-reported questionnaire that evaluates pain, stiffness, and physical function in patients with hip and knee OA. The index consists of 24 questions and the scores of the questions range from 0 (none) to 4 (very severe) and the results are evaluated over 100 points (minimum score:0 and the maximum score:100). Higher scores indicate worst knee functions.
Quality of life measure | 6 weeks
  Short form-36 will be used for quality of life assessment. SF-36 is a patient-reported questionnaire developed and made available to determine health-related quality of life. SF-36 consists of 36 items that measure eight dimensions of physical function, social function, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy/vitality, pain and general health perception. The subscales assess health between 0 and 100, with 0 showing bad health and 100 showing better health. Higher scores indicate better quality of life.
40 m fast-paced walk test | 6 weeks
  Patients will be asked to walk along the 10-meter track as fast as possible, turn around the cone at the finish, and complete the 40-meter total distance. After the patient passed the baseline in the last stage, the time will be stopped and the total time will be recorded. Lower walking distance indicates better walking capacity.
Sit-to-stand test | 6 weeks
  The patient will be seated in the middle of a chair with a height of standard 44 cm, with his back straight, arms crossed in front of his chest, and feet on the ground. The patient will be asked to get up from the chair and sit down as much as the patient could for 30 seconds. The exact number of starts will be made formed from the patient's score. Higher scores indicate better overall strength.
Stair climbing test | 6 weeks
  The patient will be asked to climb and descend the 9-step 16-20 centimetre ladder as quickly but safely as possible. The patient will be allowed to use a handrail or a walking aid, and the method used was recorded. The test will start with the start command and the time stopped when the patient returned to the starting place. The patient will be allowed to stop and rest when requested, but the duration will be continued. The total time was recorded as a score. Lower scores indicate better knee functions.
Timed up and go test | 6 weeks
  Timed up and go test (TUG) is a measurement that evaluates functional mobility, dynamic balance, fall risk and postural stability, which can be applied for different purposes in different age and patient groups. The activities that make up the test evaluate the transition from sitting to standing position, walking, turning, and sitting again, which are necessary for functional mobility and dynamic balance. The TUG test measures the time it takes an individual to get up from a standard chair with armrests and walk a distance of 3 meters, return from a designated or marked place, return to the chair, and sit down again. Lower scores indicate better mobility and balance.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Bayrak, Principal Investigator — Pamukkale University
Locations (1):
- Gökhan Bayrak, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson AW, Myrer JW, Hunter I, Feland JB, Hopkins JT, Draper DO, Eggett D. Whole-body vibration strengthening compared to traditional strengthening during physical therapy in individuals with total knee arthroplasty. Physiother Theory Pract. 2010 May;26(4):215-25. doi: 10.3109/09593980902967196. PMID 20397856
- [Background] Hsiao YH, Chien SH, Tu HP, Fu JC, Tsai ST, Chen YS, Chen YJ, Chen CH. Early Post-Operative Intervention of Whole-Body Vibration in Patients After Total Knee Arthroplasty: A Pilot Study. J Clin Med. 2019 Nov 7;8(11):1902. doi: 10.3390/jcm8111902. PMID 31703305
- [Background] Bily W, Franz C, Trimmel L, Loefler S, Cvecka J, Zampieri S, Kasche W, Sarabon N, Zenz P, Kern H. Effects of Leg-Press Training With Moderate Vibration on Muscle Strength, Pain, and Function After Total Knee Arthroplasty: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 Jun;97(6):857-65. doi: 10.1016/j.apmr.2015.12.015. Epub 2016 Jan 4. PMID 26763947
- [Background] Wang P, Yang X, Yang Y, Yang L, Zhou Y, Liu C, Reinhardt JD, He C. Effects of whole body vibration on pain, stiffness and physical functions in patients with knee osteoarthritis: a systematic review and meta-analysis. Clin Rehabil. 2015 Oct;29(10):939-51. doi: 10.1177/0269215514564895. Epub 2014 Dec 18. PMID 25525066